CLINICAL TRIAL: NCT04490473
Title: Turkish Validity And Reliability of the SARS-CoV-2 Anxiety Scale
Brief Title: Turkish of the SARS-CoV-2 Anxiety Scale
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DILEK SAYIK (Other)
Responsible Party: Sponsor-Investigator, DILEK SAYIK, Principal Investigator, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DSAYIK2; Ayfer AÇIKGÖZ (Other: ESKİŞEHİR OSMANGAZİ ÜNİVERSİTESİ); ERTUĞRUL ÇOLAK (Other: ESKİŞEHİR OSMANGAZİ ÜNİVERSİTESİ); DENİZ YİĞİT (Other: ESKİŞEHİR OSMANGAZİ ÜNİVERSİTESİ); ÖZLEM MUMCU (Other: ESKİŞEHİR ŞEHİR HASTANESİ)
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Anxiety; SARS-CoV Infection
Keywords: Coronavirus Anxiety Scale; COVID-19; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: This research will be conducted in a methodological manner in order to conduct the validity and reliability studies of the Coronary Virus Anxiety Scale in Turkish.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteer group (Other): Only volunteer participants will be included in the research. Survey forms will be sent to individuals online. Individuals who agree to participate in the study will fill in the questionnaire and send it back online.
  Interventions: Other: survey work

INTERVENTIONS:
Other: survey work — Survey forms will be sent to individuals online. Information about the study will be given to individuals with the informative text at the beginning of the questionnaire form. Individuals who agree to participate in the study will fill in the questionnaire and send it back online.

SUMMARY:
The coronavirus outbreak has adversely affected individuals in the community, as in the rest of the world. However, in order to carry out this epidemic period in a healthy and conscious manner, determining the anxiety levels of individuals in the society and supporting them psychologically is of great importance. In order to achieve this, healthcare professionals working clinically or academically have important duties. This study was planned to test its validity and reliability in order to adapt the Coronavirus Anxiety Scale to Turkish.

DETAILED DESCRIPTION:
Coronaviruses can be seen in animals and humans as infections that can be mild and severe in society. The SARS-CoV-2 virus, a type of coronavirus, started in China in December 2019 and has spread worldwide as of January 2020. The absence of vaccine and treatment for SARS-CoV-2 disease threatens health worldwide and significantly affects people's daily routine. In China, where the pandemic started, shopping malls and schools were closed for a while, and city entrances and exits were stopped for a while. Although there are similar practices in excellence, as in many countries, measures such as curfew, nursery and school closure continue to be taken for under-20s and over-65s. . The coronavirus epidemic that affects our entire life is not fully known about the disease process, WHO is defined as the pandemic of the epidemic, the nearest contact is the greatest risk of transmission, and the loss of many lives during this process affects all individuals in the society negatively and increases the level of anxiety .

It is a psychological reaction involving many emotions such as anxiety, stress, or anxiety, fear and distress that arise in a situation that threatens the safety of the individual. Conditions such as uncertainty, various diseases (cancer, epidemic, etc.) and losing a relative can cause anxiety. Outbreaks that occur suddenly and are at risk of death are among these reasons.

ELIGIBILITY:
inclusion criteria;

* individuals agree to participate in the study
* 18 years old,
* Lack of visual obstacle,
* Knowing how to speak, read and write in Turkish.

Exclusion criteria;

* individuals refuse to participate in the study
* 18 years old,
* Visually impaired,
* Does not know how to speak, read and write in Turkish

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-03-24 (Estimated); Study Completion 2021-04-24 (Estimated)

PRIMARY OUTCOMES:
Anxiety in SARS-CoV-2 | 4 weeks
  anxiety increase in SARS-CoV-2 in humans.
Ratio of SARS-CoV-2 anxiety scale to beck anxiety scale | 4 weeks
  The ratio of SARS-CoV-2 anxiety scale to beck anxiety scale is similar.

CONTACTS AND LOCATIONS:
Overall Officials: DILEK SAYIK, Principal Investigator — ESKISEHIR OSMANGAZI UNIVERSTY
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is planned to be published in the journal after the study is completed. The study will be shared with other researchers after it is published in the journal.
Supporting Information: Study Protocol
Time Frame: will be shared after the work is finished.
Access Criteria: It will be shared with researchers who want to use the anxiety scale.

REFERENCES:
- [Background] Benli, S. S., & Yıldırım, A. (2017). Hemşirelerde yaşam doyumu ve ölüme karşı tutum arasındaki ilişki. Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi, 6(4), 167-179
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Chen P, Mao L, Nassis GP, Harmer P, Ainsworth BE, Li F. Coronavirus disease (COVID-19): The need to maintain regular physical activity while taking precautions. J Sport Health Sci. 2020 Mar;9(2):103-104. doi: 10.1016/j.jshs.2020.02.001. Epub 2020 Feb 4. No abstract available. PMID 32099716
- [Background] Chen Y, Liu Q, Guo D. Emerging coronaviruses: Genome structure, replication, and pathogenesis. J Med Virol. 2020 Apr;92(4):418-423. doi: 10.1002/jmv.25681. Epub 2020 Feb 7. PMID 31967327
- [Background] Faraji A, Karimi M, Azizi SM, Janatolmakan M, Khatony A. Occupational stress and its related demographic factors among Iranian CCU nurses: a cross-sectional study. BMC Res Notes. 2019 Sep 27;12(1):634. doi: 10.1186/s13104-019-4674-5. PMID 31558161
- [Background] Lee SA. Coronavirus Anxiety Scale: A brief mental health screener for COVID-19 related anxiety. Death Stud. 2020;44(7):393-401. doi: 10.1080/07481187.2020.1748481. Epub 2020 Apr 16. PMID 32299304